CLINICAL TRIAL: NCT06076330
Title: Efficacy of 5% Albumin v/s Plasmalyte in Combination With 20% Albumin for Fluid Resuscitation in Cirrhosis With Sepsis Induced Hypotension: A Randomized Controlled Trial (ALPS Plus)
Brief Title: Efficacy of 5% Albumin v/s Plasmalyte in Combination With 20% Albumin for Fluid Resuscitation in Cirrhosis With Sepsis Induced Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-64
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Albumins; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% albumin infusion with plasmalyte (Experimental): * Plamalyte will be given at an initial bolus of 15-20 ml/kg over 15-30 mins followed by 100ml/hr maintenance
  * S. albumin > 3 g/dl: 20g of 20% iv albumin @10-15 ml/hr
  * S. albumin < 3 g/dl: 40g of 20% iv albumin @10-15 ml/hr
  Interventions: Biological: 20% Albumin; Drug: Plasmalyte
- 5% albumin at an initial bolus of 5ml/kg iv over 15-30 mins followed by 50ml/hr maintenance dose (Active Comparator): 5% albumin at an initial bolus of 5ml/kg iv over 15-30 mins followed by 50ml/hr maintenance dose
  * In case of failure to attain a sustained MAP >65 mmHg, Fluid boluses will be administered guided by lung ultrasound and IVC
  * Group A: Plasmalyte bolus of 15-20 ml/kg over 15-30 mins
  * Group B: 5ml/kg of 5% albumin over 15-30 mins
  Interventions: Biological: 5% Albumin

INTERVENTIONS:
Biological: 20% Albumin — S. albumin > 3 g/dl: 20g of 20% iv albumin @10-15 ml/hr S. albumin < 3 g/dl: 40g of 20% iv albumin @10-15 ml/hr
  Arms: 20% albumin infusion with plasmalyte
Biological: 5% Albumin — 5% albumin at an initial bolus of 5ml/kg iv over 15-30 mins followed by 50ml/hr maintenance dose In case of failure to attain a sustained MAP >65 mmHg, Fluid boluses will be administered guided by lung ultrasound and IVC.
  Arms: 5% albumin at an initial bolus of 5ml/kg iv over 15-30 mins followed by 50ml/hr maintenance dose
Drug: Plasmalyte — Plamalyte will be given at an initial bolus of 15-20 ml/kg over 15-30 mins followed by 100ml/hr maintenance
  Arms: 20% albumin infusion with plasmalyte

SUMMARY:
Cirrhotic patients with sepsis represent a very sick subset of patients and septic shock in such patients is associated with high mortality. Early initiation of intravenous fluids and antibiotics is the key to management in these patients. The choice of fluid in cirrhotic patients with sepsis induced hypotension has been studied in the past. The choice of fluid, crystalloid vs colloid, for resuscitation in such patients has been a matter of debate. In the previous study, the ALPS trial, 20% albumin use was associated with a better reversal of hypotension but was associated with an increased incidence of pulmonary complications and 5% albumin was better when compared to normal saline(FRISC study) for fluid resuscitation. No study in the past has evaluated 5% albumin against 20% albumin in combination with crystalloid. Investigator aim to study the efficacy and safety of 20% albumin with plasmalyte against 5 % albumin for fluid resuscitation in cirrhotic patients with sepsis induced hypotension.

DETAILED DESCRIPTION:
Hypothesis: Combination of 20% albumin with plasmalyte could be better than 5% albumin for fluid resuscitation in critically ill cirrhosis patients due to less incidence of hyperchloremic metabolic acidosis, dyselectrolytemia, fluid overload, and due to its cost effectiveness.

Aim: To compare the efficacy and safety of 20% albumin plus plasmalyte against 5% albumin for reversal of sepsis induced hypotension at 3 hrs in cirrhosis patients

Primary objective: To compare the efficacy of 20% albumin combined with plasmalyte against 5% albumin for reversal of shock at 3 hours after initiation of fluids in cirrhosis patients with sepsis induced hypotension

Secondary objectives:

* To study the effects of 5% albumin against 20% albumin plus plasmalyte on reversal of shock at 6, 12, 24hrs.
* to study the effects of 5% albumin against 20% albumin plus plasmalyte on arterial lactates
* To study the effect on AKI, chloride levels and coagulation in the two arms
* To study the time to initiation of noradrenaline in the two arms and the cumulative dose of norepinephrine administered in the two arms
* To study the effects of fluid resuscitation on urine output and heart rate in the two arms
* To study the effects of 5% albumin against 20% albumin plus plasmalyte on cardiopulmonary status using point of care ultrasound(POCUS)
* To study the effect of 5% albumin compared to 20% albumin plus plasmalyte on 28-day mortality.
* To study the effect of 5% albumin compared to 20% albumin plus plasmalyte on requirement and initiation of RRT
* To study the adverse effects of albumin infusion and 20% albumin plus plasmalyte infusion when used as resuscitation fluids
* To study the effect of fluid resuscitation on S. albumin concentration and effective albumin concentration in the two arms

Methodology:

Study population:

* Age - 18-75 yrs of age
* Cirrhotic patients with sepsis induced hypotension defined as mean arterial pressure less than 65mm of Hg with suspected (as per history and examination) or documented evidence of infection.

Study design: Monocentric open label randomised controlled study. The study will be conducted in Department of Hepatology, ILBS.

Study period: 1 year

Sample size: Based on the previous studies on 5% albumin and 20% albumin on fluid resuscitation, assuming that the reversal rate is approximately 11% with 5% Albumin, and 40% with 20% Albumin plus plasmalyte with alpha 5 and power 90. Investigator need to enrol 106 cases, with further 10% dropouts, it is decided to enrol 120 cases, i.e., 60 in each arm allocated randomly by block randomization method taking a block size of 10. Patients will be evaluated in ER for cirrhosis and sepsis induced hypotension

Intervention Patients after screening for all exclusion criteria will be randomised into 2 arms (group-1, receiving combination of 20% Albumin and plasmalyte) and (group-2, receiving 5% Albumin) in a ratio 1:1

* Group 1 - 20% albumin infusion with plasmalyte
* Plamalyte will be given at an initial bolus of 15-20 ml/kg over 15-30 mins followed by 100ml/hr maintenance
* S. albumin > 3 g/dl: 20g of 20% iv albumin @10-15 ml/hr
* S. albumin < 3 g/dl: 40g of 20% iv albumin @10-15 ml/hr
* Group 2 - 5% albumin at an initial bolus of 5ml/kg iv over 15-30 mins followed by 50ml/hr maintenance dose
* In case of failure to attain a sustained MAP >65 mmHg, Fluid boluses will be administered guided by lung ultrasound and IVC
* Group A: Plasmalyte bolus of 15-20 ml/kg over 15-30 mins
* Group B: 5ml/kg of 5% albumin over 15-30 mins
* Lung ultrasound and IVC will be performed at baseline and at hrly intervals for 3 hours and subsequently at 6hrly intervals for 1 day
* Fluid boluses will be administered based on the IVC and lung ultrasound - (IVC < 15)
* IVCCI>40%, and
* A profile on lung ultrasound
* Threshold(stopping rule) for fluid boluses (IVC >25)
* IVCCI <40%, or
* B profile on lung ultrasound
* Reversal of shock

Monitoring and assessment Both the groups will undergo baseline investigations including CBC, KFT, LFT, INR, Chest Xray Urine routine and microscopy, sepsis screening including blood culture, urine culture, procalcitonin, ROTEM analysis, ABG analysis, baseline 2decho, ECG, MAP, Heart rate and urine output will be monitored hourly until the reversal of shock.

Arterial lactate will be measured at 0 hours, and 3, 6, 12, 24 and 48 hours post-intervention, lactate clearance will be calculated as ([lactate initial - lactate delayed]/[lactate initial] x 100%).

IAP will be measured at baseline and at 6 hourly intervals Reversal of shock - sustained increase in MAP above 65 mmHg without the use of vasopressors.

In case of failure to attain a sustained MAP >65 mmHg, Fluid boluses will be administered guided by lung ultrasound and IVC Patients who did not attain MAP >65 mmHg after the 3 hours or with non responsiveness to fluid boluses will be initiated on vasopressors. Norepinephrine will be commenced at a rate of 7.5 µg/kg/min and gradually increased to a maximum dose of 60 µg/kg/min. Cumulative dose of norepinephrine will be recorded The patients unable to maintain a MAP of more than 65 mmHg despite the highest amount of the single vasopressor will be assigned to salvage therapy. The salvage therapy will included a combination of norepinephrine with another vasopressor (either terlipressin or vasopressin) and low dose hydrocortisone.

Same fluid will be continued in each group for 24 hours. In maintenance doses, 5% albumin will be given at a maintenance dose of 50ml/hr in 5% albumin group and plasmalyte at 100ml/hr in combination arm. Cumulative fluid administered in both groups will be recorded.

Antibiotics will be initiated on an empirical basis as per our institute's microbiological epidemiology and will be revised, if necessary, based on culture positivity.

Electrolyte correction will be given as per the requirement Enteral or parenteral nutrition depending upon tolerance will be initiated. Anti-coma measures will be given for hepatic encephalopathy and RRT for standard renal indications which will include metabolic acidosis, fluid overload, hyperkalemia, and advanced uremia Time to initiation of RRT for both groups will be recorded.

Lung ultrasound and IVC will be performed at baseline and at hrly intervals for 3 hours and subsequently at 6hrly intervals for 1 day Fluid boluses will be administered based on the IVC and lung ultrasound - IVC < 15 IVCCI>40%(spontaneously breathing patients) and IVCDI>18%(Mechanically ventilated patients), and A profile on lung ultrasound Threshold(stopping rule) for fluid boluses (IVC >25) IVCCI <40% in spontaneously breathing patients and IVCDI<18% in mechanically ventilated patients, or B profile on lung ultrasound

Stopping rule:

* Development of adverse effects
* Need for 2nd vasopressor

STATISTICAL ANALYSIS: Continuous data- Student's t test

* Nonparametric analysis- Mann Whitney test
* Survival outcome By Kaplan-Meier method curve.
* For all tests, p≤ 0.05 will be considered statistically significant.
* Analysis will be performed using SPSS.
* The analysis will be done with intention to treat and per protocol analysis if applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Age - 18-75 yrs of age
2. Cirrhotic patients with sepsis induced hypotension defined as mean arterial pressure less than 65mm of Hg with suspected (as per history and examination) or documented evidence of infection.

Exclusion Criteria:

1. Patients with other causes of hypotension
2. Patients who have already received bolus of 5% albumin or plasmalyte or >2L of fluids
3. Patients with structural heart disease or known diastolic dysfunction or cirrhotic cardiomyopathy
4. Patients who are on vasopressors or inotropes,
5. Patients already receiving renal replacement therapy
6. Patients with known chronic obstructive lung disease or congestive heart failure
7. Patients with serum albumin below 1.5 g/dl
8. Patients in need of surgical intervention
9. Pregnant or lactating women
10. Patients with a previous adverse reaction to human albumin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving Mean Arterial Pressure above 65mm of Hg at 3 hrs after intervention | 3 hours

SECONDARY OUTCOMES:
Proportion of patients with reversal of shock in the two groups. | 6 hours
Proportion of patients with reversal of shock in the two groups. | 12 hours
Proportion of patients with reversal of shock in the two groups. | 24 hours
Effect of fluid resuscitation on lactate clearance in the two groups. | 0 hour
Effect of fluid resuscitation on lactate clearance in the two groups. | 1 hour
Effect of fluid resuscitation on lactate clearance in the two groups. | 3 hour
Effect of fluid resuscitation on lactate clearance in the two groups. | 6 hour
Effect of fluid resuscitation on lactate clearance in the two groups. | 12 hour
Effect of fluid resuscitation on lactate clearance in the two groups. | 24 hour
Cumulative amount of fluid used in two arms. | 24 hour
Time to initiation of norepinephrine in the two arms | 24 hour
Cumulative dose of norepinephrine in two arms | 24 hour
Length of ICU stay in the two groups | 28 days
Mortality in the two groups | 28 days
To study the adverse effects (including pulmonary, metabolic and coagulopathy) in the two groups. | Day 1
To study the adverse effects (including pulmonary, metabolic and coagulopathy) in the two groups. | Day 3
To study the adverse effects (including pulmonary, metabolic and coagulopathy) in the two groups. | Day 7
To study the adverse effects (including pulmonary, metabolic and coagulopathy) in the two groups. | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India